CLINICAL TRIAL: NCT06003543
Title: The Effect of Virtual Reality Application on Pain, Fear and Anxiety in Patients Undergoing Colonoscopy:
Brief Title: The Effect of Virtual Reality Application on Pain, Fear and Anxiety in Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-19003918-730.08.03-347141
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality
Keywords: Fear; Colonoscopy,; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): virtual glasses will be applied
  Interventions: Behavioral: Virtual Reality
- Control (No Intervention): no application will be made

INTERVENTIONS:
Behavioral: Virtual Reality — Virtual Reality
  Arms: Virtual Reality

SUMMARY:
Colonoscopy; It is a method that allows viewing the large intestines and diagnosing or treating gastrointestinal system diseases by entering through the anus with a flexible, thin tube with a camera at the end, called a colonoscope. All parts of the large intestine with colonoscopy; ascending colon, hepatic flexure, transverse colon, splenic flexure, descending colon, sigmoid colon, rectum and anal canal by retroflexion can be evaluated. Colonoscopic interventions applied in gastroenterology cause pain, fear and anxiety in patients.

DETAILED DESCRIPTION:
High anxiety levels before the procedure can negatively affect the procedure by reducing patient compliance and may lead to the incompleteness of the procedure. Anxiety and fear experienced during colonoscopy cause more pain during the procedure.

In addition to pharmacological methods, there are non-pharmacological methods to provide patient comfort and manage the level of pain, fear and anxiety in interventional procedures such as colonoscopy. The methods used can be grouped under three main headings: physical, supportive and cognitive-behavioral. Cognitive-behavioral methods, which can be performed with practices such as relaxation and distraction, help control pain, fear and anxiety level.

The virtual reality application, developed thanks to the advancement of computer technology, is used as a cognitive-behavioral method to alleviate pain, fear and anxiety. With this method, the process of processing incoming pain signals slows down in patients who focus their attention on the environment they see, and fear, anxiety and pain are perceived less. It is important to relieve the patient's pain, fear and anxiety before colonoscopic interventions, to diagnose the patient correctly, to facilitate the health personnel who will perform the procedure, to facilitate the patient's compliance with the procedure, to prevent possible complications and to increase patient satisfaction. This study was planned to examine the effect of relaxation exercise, which will be performed with virtual reality application, which will distract their attention before and during the colonoscopy, on the experienced pain, fear and anxiety levels.

The research will be conducted as a randomized, experimental study with a pretest-posttest control group. The sample of the study will be composed of a total of 46 patients, 23 experimental and 23 control groups, who will be subjected to colonoscopy between August 2023- August 2024 in the Colonoscopy Unit of the Gastroenterology Polyclinic of Fırat University Hospital. Virtual reality application will be applied to the patient in the experimental group by the researcher 10 minutes before the procedure and 10-15 minutes during the procedure. The first measurement will be obtained by applying the Visual Analog Scale-Pain, Visual Analog Scale-Fear, Visual Analog Scale-Anxiety, State-Trait Anxiety Inventory (DSQ) and Patient Information Form to the patient in the experimental group before the procedure. The second measurement will be obtained by applying the Visual Analog Scale-Pain, Visual Analog Scale-Fear, Visual Analog Scale-Anxiety and State-Trait Anxiety Scale (DSQ) to the patient 10-15 minutes after the procedure. No intervention will be performed on the patients in the control group. 1 measurement will be obtained by applying the Patient Information Form, Visual Analog Scale-Pain, Visual Analog Scale-Fear, Visual Analog Scale-Anxiety and State-Trait Anxiety Scale before the procedure only. After the procedure, the second measurement will be obtained by re-applying the other forms except the Patient Information Form. The data will be analyzed using the SPSS 23 program. Shapiro Wilk test, t test, Mann-Whitney U test, Wilcoxon test and Chi-square analysis will be used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish
* Having cognitive competence to answer data collection tools
* Absence of communication problems (hearing, language, understanding, etc.)
* Not having a psychiatric diagnosis
* Absence of a history of convulsions
* Patients who underwent local application in colonoscopy

Exclusion Criteria:

* Those with communication problems
* Those with psychiatric problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale -Pain | 1 hours later
  Patients are asked to show the intensity of pain on a 10 cm long vertical or horizontal line during activity or rest. It has numbered shapes ranging from 1-10. The line has 0 at the beginning and 10 at the end. 10 means unbearable pain, 0 means no pain. The VAS scale is frequently used in the evaluation of pain severity. While the patient marks the pain he/she has felt on this line, each point marked is measured in cm
Visual Analog Scale - Fear | 1 hours later
  Patients are asked to show the intensity of fear on a 10 cm long vertical or horizontal line during activity or rest. It has numbered shapes ranging from 1-10. The line has 0 at the beginning and 10 at the end. 10 means unbearable fear, 0 means no fear. The VAS scale is frequently used in the evaluation of fear severity. While the patient marks the fear he/she has felt on this line, each marked point is measured in cm
Visual Analog Scale -Anxiety | 1 hours later
  Patients are asked to show the intensity of anxiety on a 10 cm long horizontal line during activity or rest. The line has 0 at the beginning and 10 at the end. 10 means unbearable pain, 0 means no pain. VAS is frequently used in the evaluation of pain intensity. While the patient marks the anxiety he/she has felt on this line, each marked point is measured in cm
State-Trait Anxiety Inventory | 1 hours later
  Developed by Spielberg et al. (1970) to measure the state and trait anxiety levels of individuals, the scale, which consists of two parts and the English name is Speilberg's State-Trait Anxiety Inventory (STAI), is a self-tested reliability and validity study in Turkish by Öner and Le Compte (1977). assessment scale (37-38) In this study, the part of the scale measuring trait anxiety was used to determine the trait anxiety levels of the patients. Trait Anxiety Inventory is a 4-point Likert-type with 20 items and is scored as "never": 1, "a little": 2, "a lot": 3, "completely": 4, according to the severity of the feelings, thoughts or behaviors expressed by the items. . There are direct or reverse scored statements in the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan B.TURAN, Principal Investigator — Firat University
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No